CLINICAL TRIAL: NCT06853847
Title: Effect of Position Change on Pain, Comfort and Vascular Complications After Coronary Angiography: A Double-Blind Randomized Controlled Trial
Brief Title: Effect of Position Change on Pain, Comfort and Vascular Complications After Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Assistant Professor of Nursing, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0005
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Angiopathy, Peripheral; Pain
MeSH Terms: conditions — Peripheral Vascular Diseases; Pain

STUDY DESIGN:
Intervention Model Description: This study is a double-blind randomized controlled trial planned to investigate the effect of position change after coronary angiography on pain, comfort and vascular complications.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be divided into experimental and control groups. Patients will know that they are participating in the study and the interventions that will be applied to them, but they will be blinded by not knowing which group they are in. The study data will be collected by a second researcher who is blinded to the groups. In the statistical analysis of the data, the groups will be labeled as group 1 and group 2, and the third researcher will be blinded when evaluating the results. Thus, the third researcher will be blinded to the study groups. In order to avoid bias in the evaluation of the results, the first researcher who is not blinded will not participate in any stage of the evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- back position group (Experimental): The bed levels of the patients in the experimental group changed the patient's position every 2 hours immediately after catheter removal and sandbag placement in the following order: supine position with a 15° head angle, semi-Fowler position with a 30° head angle, and lateral right or left position with a 15° head angle.
  Interventions: Other: The bed levels of the patients in the experimental group changed the patient's position
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: The bed levels of the patients in the experimental group changed the patient's position — The bed levels of the patients in the experimental group changed the patient's position
  Arms: back position group

SUMMARY:
Today, complementary and alternative treatments are frequently used to maintain health and well-being, reduce symptoms of diseases, and provide relaxation. Nurses contribute to the healing process by using pharmacological and nonpharmacological methods. Pharmacological methods cause nausea, vomiting, respiratory depression, gastrointestinal and urinary system complications in individuals. Therefore, nonpharmacological methods without side effects are gaining importance. Nonpharmacological methods are easy and simple nursing interventions that do not have side effects, are cost-effective, can be easily taught to the patient, reduce pain and anxiety. They can also be used in addition to pharmacological methods and are preferred in patients who do not take medication or are unwilling to take medication. Providing a safe position without vascular complications and back pain after the procedure is very important for both the patient and the nurse who cares for the patient. Existing studies on post-intervention position changes have reported low incidences of bleeding and back pain, resulting in higher levels of patient comfort and satisfaction. These studies evaluated different angles of elevating the head of the bed and recommended further studies to evaluate the possibility of shifting patients to other positions after transfemoral cardiac interventions.

DETAILED DESCRIPTION:
Therefore, the aim of this study was to investigate the effect of position change after coronary angiography on pain, comfort and vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

  * Agree to participate in the study
  * Not undergoing emergency coronary angiography
  * Not consuming coffee or hypnotic drugs at least 12 hours ago
  * No history of chronic pain (e.g. arthritis)
  * Not addicted to alcohol or drugs
  * No psychological problems (such as depression, anxiety disorder)
  * Not using anxiolytics

Exclusion Criteria:

* • Not willing to participate in the study

  * Developing delirium during the follow-up period
  * Developing complications after coronary angiography (such as bleeding etc.)
  * Arrhythmia
  * Hemodynamic instability
  * Hereditary bleeding disorders
  * Platelet count less than 100,000/mm3
  * Abnormal coagulation parameters (high INR and/or aPTT)
  * History of percutaneous coronary intervention (PCI)
  * Multiple or bilateral punctures in the femoral artery
  * Presence of hematoma on arrival after the procedure
  * Radial access
  * Bleeding at the access site or at the access dressing site
  * Body mass index (BMI) ≥ 35 kg/m2
  * Back pain before treatment
  * Patients with spinal cord disease
  * Patients with vertebral disc disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Average Pain Score on Visual Analog Scale (VAS) | 0 hour (baseline), 1st hour, 2nd hour, 3rd hour
  Pain will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (severe pain). Higher scores indicate more severe pain.
Average Score on Immobilization Comfort Scale (ICS) | 0 hour (baseline), 1st hour, 2nd hour, 3rd hour
  Comfort during immobilization will be measured using the Immobilization Comfort Scale (ICS), a 20-item Likert-type scale ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate greater comfort. Cronbach's alpha in this study ranged from 0.77 to 0.84.
Vascular Complication Score | 0 hour (baseline), 1st hour, 2nd hour, 3rd hour
  Vascular complications will be assessed using the Oozing and Bleeding Scale and the Ecchymosis and Hematoma Formation Scale developed by Elsaman (2022). Categories include: no bleeding/ecchymosis/hematoma, oozing/bleeding <2 cm², bleeding ≥2 cm², ecchymosis <2 cm², hematoma ≥2 cm². Higher scores indicate more severe vascular complications.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu NAL, PhD, Study Director — Kütahya Health Sciences University, Faculty of Health Sciences; Mehmet Ali ASTARCIOĞLU, Prof., Study Director — Kütahya Health Sciences University, Faculty of Health Sciences
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No